CLINICAL TRIAL: NCT00806910
Title: Evaluation of the Diuretic and Renal Effects of Vaprisol When Administered Along With Furosemide and Nesiritide Continuous Infusion
Brief Title: Diuretic and Renal Effects of Vaprisol When Administered Along With Furosemide and Nesiritide Continuous Infusion
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor support withdrawn
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Darshak H. Karia, MD. Director, Heart Failure Services, Albert Einstein Heart and Vascular, Albert Einstein Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HN-4040
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; conivaptan; Diuresis
MeSH Terms: conditions — Heart Failure | interventions — conivaptan; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Subjects will be treated with Intravenous Vaprisol along with Nesiritide infusion and intravenous Furosemide (either continuous infusion or bolus injections - total dose of Furosemide received will be calculated at the end of the study).
  Interventions: Drug: Conivaptan
- Placebo (Placebo Comparator): Subjects will be given Placebo (at the same rate of Vaprisol given in the treatment arm) along with Nesiritide infusion and intravenous Furosemide (either continuous infusion or bolus injections - total dose of Furosemide received will be calculated at the end of the study).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Conivaptan — IV Vaprisol initially at 20 mg IV injection over 30 minutes, followed by a 20 mg IV infusion over the next 24 hours (i.e. 20 mg bolus, 20 mg continuous infusion approximately 24 hrs).
  Other Names: Vaprisol
  Arms: Treatment
Other: Placebo — Placebo (will be given at the same rate of Vaprisol given in the treatment arm)
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Heart Failure is a growing and challenging public health concern in the United States. Heart failure commonly manifests as a syndrome of salt and water retention. Arginine vasopressin is a peptide hormone that is intimately involved in salt and water homeostasis. AVP is released into the circulation in response low blood volume and hypernatraemia. Despite fluid overload, vasopressin levels are often inappropriately elevated in patients with heart failure and LV dysfunction. Data suggest that vasopressin may also contribute to the deleterious circulatory response in patients with heart failure and play a role in the development and progression of the disease process. In their study, Udelson et al. showed that vasopressin receptor antagonism with Conivaptan resulted in significant diuresis with stable hemodynamics in advanced heart failure patients. Currently Intravenous diuretics and vasodilators are the standard of care in treating patients with acute decompensated heart failure. We will be studying the renal and diuretic effects of add on therapy with intravenous Conivaptan in patients receiving intravenous Nesiritide and intravenous diuretics.

DETAILED DESCRIPTION:
Heart failure effects 5 to 6 million Americans and is increasing in prevalence. There are about 550, 000 new cases of heart failure every year and about 3 million admissions for acute decompensated heart failure every year. The total cost of heat failure on the health systems is upwards of 35 billion dollars per year. Despite advances in medical care, the hospital readmission rate is 20% at one month and 50% at six months. This prevailing situation mandates further exploration of novel therapeutic targets to treat this complex disease.

Vasopressin levels are often elevated in patients with heart failure and LV dysfunction which is paradoxical and inappropriate. It has been hypothesized that high levels of circulating vasopressin may play an important role not only in the pathophysiology of the heart failure syndrome but also contribute to its disease progression.

Studies have shown that Conivaptan, a Vasopressin antagonist results in favorable changes in hemodynamics and urine output without affecting blood pressure or heart rate. No consensus has been reached for Conivaptan to be used as a sole agent in Acute Decompensated Heart Failure (ADHF) patients and IV loop diuretics and/or vasodilators such as Nesiritide are used as the prime treatment for vascular congestion. This prevailing situation brings the questions whether, Conivaptan can be used as an adjunct to IV Furosemide and/or Nesiritide presenting with ADHF.We intend to investigate this question in a cohort of heart failure patients with hyponatremia.

This study will enroll 60 patients ( who meets all the inclusion criteria and none of the exclusion criteria), admitted to the Albert Einstein Medical Center with the diagnosis of Acute Decompensated Heart Failure (New York Heart Association class 3 and 4). The study population will be divided into 2 groups; a treatment group and a placebo group as described below. Each group will be comprised of 30 patients.

The treatment group will be treated with Nesiritide infusion, intravenous Furosemide (either continuous infusion or bolus injection- total dose of Furosemide received at the end of the study will be calculated) and IV Vaprisol. The placebo group will be given Nesiritide infusion and intravenous Furosemide(either continuous infusion or bolus injection) and placebo. Treatment will be continued in both groups for 24-36 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 and able to consent
* LVEF ≤40% (as measured within last 6 months before entering into the study)
* Patients with Acute Decompensated Heart Failure (ADHF) (NYHA class 3 & 4)
* Patients with estimated GFR >40ml/min as calculated by Cockcroft-Gault or MDRD formula
* Serum Sodium level <135 meq/L
* Ability to understand and willing to sign informed consent
* Willingness to follow-up in the clinic as outpatient

Exclusion Criteria:

* Patients with Acute Coronary Syndrome (ACS: Unstable angina, NSTEMI or STEMI)
* Patients on pressors (including Vasopressin analogs) for hemodynamic stability
* Supine systolic blood pressure <100 mm Hg
* Hypersensitivity to Conivaptan
* Concomitant use of medications that affects hepatic drug metabolism (e.g. Ketoconazole, Itraconazole, Ritonavir, Indinavir, Clarithromycin etc.)
* Significant liver dysfunction (ALT & AST more than twice the upper limit of normal)
* Uncontrolled bradyarrhythmias or tachyarrhythmias
* Pacemaker or defibrillator implantation or other cardiac surgery <60 days
* Severe obstructive pulmonary disease
* Significant uncorrected valvular or congenital heart disease
* Obstructive cardiomyopathy
* Significant renal impairment (defined as a serum creatinine >2.5 mg/dL or creatinine clearance <40 ml/min).
* Radiocontrast infusion within <7 days
* Pregnant or lactating female subject
* Untreated severe hyperthyroidism, hypothyroidism or adrenal insufficiency
* Expected requirement for emergent treatment of hypernatremia during the course of the study
* Known urinary outflow obstruction, unless subject is, or can be catheterized during the study
* Serum albumin < 1.5 gm/dl documented any time during any time during seven days prior to study drug administration
* Any concurrent illness, which in opinion of the investigator, may interfere with treatment or evaluation of safety.
* White blood cell count (WBC) count < 3000 /mL documented any time during seven days prior to study drug administration or anticipated drop in WBC count <3000/mL during the period of study due to chemotherapy.
* Participation in another clinical trial of an investigational drug (including placebo) or device within 30 days of screening for entry into the present study
* Subject has moderate ascites on physical examination secondary to hepatic dysfunction (ascites primarily related to cardiac dysfunction will be allowed as long as subject does not have cardiac cirrhosis).
* Subject has moderate to severe hepatic impairment as evidenced by Child-Pugh B or C criteria.
* Subject has a history of hepatic encephalopathy, hematemesis or melena.
* Subjects with altered mental status due to severe hyponatremia.
* Patient belonging to a vulnerable population such as institutionalized person, prisoners and persons with decisional incapacity or dementia.
* Patients on medications which are known to cause drug interactions such as Nicardipine, lovastatin, Ritonovir, Doxorubicin Etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Degree of diuresis as measured by weight change and intake and output measurement | Post infusion, Pre discharge and at 30 day Post discharge

SECONDARY OUTCOMES:
Length of stay (LOS) in hospital | Concurrent
Clinical status based on NYHA criteria | Pre-discharge and 30-day post-discharge follow up
Serum electrolytes | Pre and Post infusion
BUN and Serum Creatinine concentration | Post infusion, Pre discharge and at 30 day Post discharge
Number of readmissions due to ADHF | Within 30-day post-discharge follow up
Dyspnea assessment by Visual Analog Scale score | Post infusion, Pre discharge and at 30 day Post discharge
Subjective feeling based on Minnesota - Living with Heart Failure Questionnaire | Pre-discharge and 30-day post-discharge follow up

CONTACTS AND LOCATIONS:
Overall Officials: Darshak H Karia, MD, Principal Investigator — Albert Einstein Medical Center